CLINICAL TRIAL: NCT04180501
Title: A Phase II Study on the Treatment of Advanced Non-small Cell Lung Cancer With Brain Metastasis by SRS Sequential Sintilimab
Brief Title: SRS Sequential Sindilimab in Brain Metastasis of NSLSC
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xiaorong Dong (Other)
Responsible Party: Sponsor-Investigator, Xiaorong Dong, Professor, Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Organization: Union Hospital, Tongji Medical College, Huazhong University of Science and Technology (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: sintilimab
Record Dates: First submitted 2019-11-12; First posted 2019-11-27 (Actual); Last update posted 2019-11-27 (Actual); Status verified 2019-11

CONDITIONS: NSCLC Stage IV; Brain Metastases; SRS; Sintilimab
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung; Brain Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SRS sequential sintilimab (Experimental)
  Interventions: Combination Product: SRS sequential sintilimab

INTERVENTIONS:
Combination Product: SRS sequential sintilimab — The subjects first received a targeted radiotherapy of SRS, and started the treatment of sintilimab per 3 weeks within 35 days after SRS.

SUMMARY:
A phase II study on the treatment of advanced non-small cell lung cancer with brain metastasis by SRS sequential sintilimab

ELIGIBILITY:
Inclusion Criteria:

* non-small cell lung cancer patients with less than brain metastases
* Patients must have received at least the first-line anti-tumor treatment, and the front-line treatment must include chemotherapy or targeted treatment with a platinum containing combination scheme, but not anti-PD-1 / L1 treatment
* Patients who have not received intracranial local treatment before

Exclusion Criteria:

* Patients who toke major surgery within 4 weeks prior to enrollment or had ununited wounds
* Patients with hemorrhage in intracranial metastasis

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Estimated)
Dates: Start 2019-11 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
iPFSof NSCLC patients receiving SRS sequential sintilimab | 1 year
  From the beginning of treatment to the end of follow-up study, when the longest diameter of brain metastases treated by SRS was more than 30% smaller than the baseline level at any time of efficacy evaluation, the objective remission of the lesions was achieved. The time from the objective remission to the next progress of the intracranial lesions was recorded as the intracranial progression-free survival(iPFS).

CONTACTS AND LOCATIONS:
Locations (1):
- Union hospital, Wuhan, Hubei, China